CLINICAL TRIAL: NCT00787852
Title: A Phase I Study of Dasatinib With Concurrent Chemoradiation for Stage III NSCLC Principal Investigator: Howard Safran, MD.
Brief Title: A Study of Dasatinib With Concurrent Chemoradiation for Stage III Non-Small Cell Lung Cancer (NSCLC)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: for efficacy and safety reasons
Sponsor: Brown University (Other)
Collaborators: Rhode Island Hospital (Other); Memorial Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, howard safran, Principal Investigator, Brown University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG-NSCL-216
Record Dates: First submitted 2008-11-07; First posted 2008-11-10 (Estimated); Results first posted 2013-09-25 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-07

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: dasatinib; radiation; paclitaxel; carboplatin; NSCLC; safety addition of dasatinib to chemo RT stage III NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1: Radiation, Paclitaxel, Carbo, Dasatinib days 1-47 (Experimental): Locally Advanced Stage III NSCLC DAY Radiation 1-5 8-12 15-19 22-26 29-33 36-40 43-47 Paclitaxel 1 8 15 22 29 36 43 Carboplatin 1 8 15 22 29 36 43 Dasatinib & Maintenance Dasatinib RT: External radiotherapy, 64.8 Gy, for 35 fx Paclitaxel: 50 mg/m2/week over 1 hour IV infusion days 1, 8, 15, 22, 29, 36, 43 Carboplatin: AUC = 2 IV infusion days 1, 8, 15, 22, 29, 36, 43
  Dasatinib is to be taken 1x daily
  1. 50 mg daily 100 mg daily
  2. 70 mg daily 100 mg daily
  3. 100 mg daily 100 mg daily
  Maintenance x 2 years*
  Interventions: Drug: Group 1: Radiation, Paclitaxel,Carbo, Dasatinib days 1-47
- Group 2: Radiation, Paclitaxel, carbo, Dasatinib days 1-38 (Experimental): Group 2: Neoadjuvant Therapy for Potentially Resectable Stage III NSCLC SCHEMA DAY Radiation 1-5 8-12 15-19 22-26 29-33 36-38 Paclitaxel 1 8 15 22 29 36 Surgery Carboplatin 1 8 15 22 29 36 Dasatinib & Maintenance Dasatinib RT: External radiotherapy 50.4 Gy, 1.8 Gy/fx for 28 fx Paclitaxel: 50 mg/m2/week over 1 hour IV infusion days 1, 8, 15, 22, 29, 36 Carboplatin: AUC = 2 IV infusion days 1, 8, 15, 22, 29, 36
  Dasatinib is to be taken 1x daily
  1. 50 mg daily 100 mg daily
  2. 70 mg daily 100 mg daily
  3. 100 mg daily 100 mg daily Maintenance x 2 years*
  Interventions: Drug: Group 2: Radiation, Paclitaxel, Carbo, Dasatinib days 1-38

INTERVENTIONS:
Drug: Group 1: Radiation, Paclitaxel,Carbo, Dasatinib days 1-47 — Locally Advanced Stage III NSCLC DAY Radiation 1-5 8-12 15-19 22-26 29-33 36-40 43-47 Paclitaxel 1 8 15 22 29 36 43 Carboplatin 1 8 15 22 29 36 43 Dasatinib & Maintenance Dasatinib RT: External radiotherapy, 64.8 Gy, for 35 fx Paclitaxel: 50 mg/m2/week over 1 hour IV infusion days 1, 8, 15, 22, 29, 36, 43 Carboplatin: AUC = 2 IV infusion days 1, 8, 15, 22, 29, 36, 43
  Dasatinib is to be taken 1x daily
  1. 50 mg daily 100 mg daily
  2. 70 mg daily 100 mg daily
  3. 100 mg daily 100 mg daily
  Maintenance x 2 years*
  Other Names: Group 1: Locally Advanced Stage III NSCLC
  Arms: Group 1: Radiation, Paclitaxel, Carbo, Dasatinib days 1-47
Drug: Group 2: Radiation, Paclitaxel, Carbo, Dasatinib days 1-38 — Group 2: Neoadjuvant Therapy for Potentially Resectable Stage III NSCLC SCHEMA DAY Radiation 1-5 8-12 15-19 22-26 29-33 36-38 Paclitaxel 1 8 15 22 29 36 Surgery Carboplatin 1 8 15 22 29 36 Dasatinib & Maintenance Dasatinib RT: External radiotherapy 50.4 Gy, 1.8 Gy/fx for 28 fx Paclitaxel: 50 mg/m2/week over 1 hour IV infusion days 1, 8, 15, 22, 29, 36 Carboplatin: AUC = 2 IV infusion days 1, 8, 15, 22, 29, 36
  Dasatinib is to be taken 1x daily
  1. 50 mg daily 100 mg daily
  2. 70 mg daily 100 mg daily
  3. 100 mg daily 100 mg daily Maintenance x 2 years*
  Other Names: Group 2: Neoadjuvant Therapy for Potentially Resectable Stage III NSCLC
  Arms: Group 2: Radiation, Paclitaxel, carbo, Dasatinib days 1-38

SUMMARY:
The purpose of this study is to evaluate if a maximum dose of 100 mg of dasatinib with concurrent chemoradiation can be tolerated in patients with chemotherapy naive stage III NSCLC in separate cohorts of locally advanced and potentially resectable disease.

DETAILED DESCRIPTION:
Describe the safety of maintenance dasatinib, 100 mg/day for 2 years, in patients with stage III NSCLC.

For patients with potentially resectable disease, to assess the pathologic complete response following neoadjuvant dasatinib, paclitaxel, carboplatin and 50.4 Gy concurrent radiation.

For patients with locally unresectable disease, to obtain radiographic response data following dasatinib, paclitaxel, carboplatin and 64.8 Gy radiation.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven (either histologic or cytologic) diagnosis of Stage IIIA or IIIB non-small cell lung cancer; excluding patients with N3 disease based on supraclavicular or contralateral hilar adenopathy, [according to AJCC Staging, 6th edition; see Appendix G] within 4 weeks of registration.
* No prior chemotherapy or radiation for lung cancer. No prior radiation for any malignancy within the radiation field.
* Patients may be potentially resectable or unresectable.
* Stage III A or B disease, including no distant metastases- based on following diagnostic workup:

  * History/physical examination prior to registration.
  * CT Scan of the chest or Pet Scan within 28 days of study entry.
  * CT Scan of abdomen or MRI of abdomen or Pet Scan within 28 days of study entry.
  * An MRI of the brain or Head CT Scan with contrast within 28 days of study entry.
  * Total body PET scan within 6 weeks of study entry is highly recommended and required for operable patients. If a PET scan is performed then a bone scan is not required.
  * A bone scan should be performed within 6 weeks of study entry. A bone scan is not needed if a PET scan is performed.
  * Mediastinoscopies are highly recommended. Mediastinoscopy is required for all patients not undergoing PET scans and for those who are operable.
* Patients must have measurable or evaluable disease.
* Patients with post-obstructive pneumonia are eligible.
* Patients must be at least 3 weeks from prior thoracotomy (if performed)
* ECOG Performance Status 0-1. Age > 18.
* Post-op predicted FEV1 > 40% to be eligible for surgical resection.
* CBC/differential obtained within 2 weeks prior to registration on study, with adequate bone marrow function defined as follows:

  * Absolute neutrophil count (ANC) > 1,500 cells/ul.
  * Platelets > 100,000 cells/ul.
  * Hemoglobin > 9.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb > g/dl is acceptable.)
  * PT, PTT all Grade 0-1
  * Serum creatinine < 1.5 x ULN
  * Total bilirubin < 2.0 times the institutional Upper Limit of Normal (ULN)
  * AST and ALT < 2.5 x the ULN
  * Serum Na, K+, Mg2+, Phosphate in normal range (LLN)
  * Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 72 hours prior to the start of study drug administration.
* Persons of reproductive potential must agree to use and utilize an adequate method of contraception throughout treatment and for at least 4 weeks after study drug is stopped prior to study enrollment, women of childbearing potential must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy.
* If you are capable of giving birth to or fathering a child, you must agree to use a form of birth control (examples of effective birth control are: a condom or a diaphragm with spermicidal jelly; oral, injectable, or implanted birth control; or abstinence) that is medically acceptable to your study doctor while taking part in this research study. This is necessary because the treatment involved in this study may be significantly teratogenic.
* PFT's within 8 weeks of study entry
* EKG within 6 weeks of study entry
* Ability to take oral medication (dasatinib must be swallowed whole)
* Patient must sign study specific informed consent prior to study entry.
* Patient agrees to discontinue St. Johns Wort while receiving dasatinib therapy (discontinue St. Johns Wort at least 5 days before starting dasatinib)

Exclusion Criteria:

* Supraclavicular disease
* Pleural or pericardial effusion of any grade
* No prior malignancy [other than the one treated in this study] which required radiotherapy or systemic treatment within the past 3 years
* Severe, active co-morbidity, defined as follows:
* Cardiac Symptoms; any of the following should be considered for exclusion:

  * Uncontrolled angina, congestive heart failure or MI within (6 months)
  * Diagnosed congenital long QT syndrome
  * Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes)
  * Prolonged QTc interval on pre-entry electrocardiogram (> 450 msec)
  * Subjects with hypokalemia or hypomagnesemia if it cannot be corrected prior to dasatinib administration
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive.
  * Protocol-specific requirements may also exclude immuno-compromised patients
  * History of significant bleeding disorder unrelated to cancer, including:
  * Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease).
  * Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies).
  * Ongoing or recent (< 3 months) significant gastrointestinal bleeding
  * Concomitant Medications, any of the following should be considered for exclusion:

    * Category I drugs that are generally accepted to have a risk of causing Torsades de Pointes including: (Patients must discontinue drug 7 days prior to starting dasatinib):

      1. quinidine, procainamide, disopyramide
      2. amiodarone, sotalol, ibutilide, dofetilide
      3. erythromycin, clarithromycin
      4. chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide, cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious) illness

  * Women who:are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 4 weeks after cessation of study drug, or have a positive pregnancy test at baseline, or are pregnant or breastfeeding
* Any history of allergic reaction to paclitaxel or other taxanes, or to carboplatin.

  * Uncontrolled neuropathy grade 2 or greater regardless of cause.
  * Patients who are on full dose aspirin, Clopidogrel bisulfate (plavix) or other GPIIb/IIIa platelet inhibitors are not eligible. Patients must have these agents stopped within 7 days of initiated treatment. Patients may be on low dose aspirin (81 mg/day).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-03; Primary Completion 2011-03 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Safran, md, Study Director — Brown University
Locations (1):
- Lifespan Hospitals, Providence, Rhode Island, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled 3/25/09 and last patient was enrolled 1/4/11. 11 patients enrolled, 10 were treated secondary to 1 patient withdrawing prior to treatment.
Groups:
- Group 1: Dasatinib 50mg: DAY Radiation 1-5 8-12 15-19 22-26 29-33 36-40 43-47 Paclitaxel 1 8 15 22 29 36 43 Carboplatin 1 8 15 22 29 36 43 Dasatinib & Maintenance Dasatinib RT: External radiotherapy, 64.8 Gy, for 35 fx Paclitaxel: 50 mg/m2/week over 1 hour IV infusion days 1, 8, 15, 22, 29, 36, 43 Carboplatin: AUC = 2 IV infusion days 1, 8, 15, 22, 29, 36, 43
  Dasatinib is to be taken 1x daily 50 mg daily
  Maintenance x 2 years*
- Group 2: Dasatinib 70mg: DAY Radiation 1-5 8-12 15-19 22-26 29-33 36-40 43-47 Paclitaxel 1 8 15 22 29 36 43 Carboplatin 1 8 15 22 29 36 43 Dasatinib & Maintenance Dasatinib RT: External radiotherapy, 64.8 Gy, for 35 fx Paclitaxel: 50 mg/m2/week over 1 hour IV infusion days 1, 8, 15, 22, 29, 36, 43 Carboplatin: AUC = 2 IV infusion days 1, 8, 15, 22, 29, 36, 43
  Dasatinib is to be taken 1x daily 70 mg daily
  Maintenance x 2 years*
Period: Overall Study
Arm/Group | Group 1: Dasatinib 50mg | Group 2: Dasatinib 70mg
Started | 6 | 5 (The study was terminated prior to enrolled to group 2)
Completed | 5 (1 patient withdrew consent prior to starting) | 5
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: 11 were enrolled but 10 were treated
Groups:
- Group 1: DAY Radiation 1-5 8-12 15-19 22-26 29-33 36-40 43-47 Paclitaxel 1 8 15 22 29 36 43 Carboplatin 1 8 15 22 29 36 43 Dasatinib ----------------------------------------------------------------------Maintenance Dasatinib RT: External radiotherapy, 64.8 Gy, for 35 fx Paclitaxel: 50 mg/m2/week over 1 hour IV infusion days 1, 8, 15, 22, 29, 36, 43 Carboplatin: AUC = 2 IV infusion days 1, 8, 15, 22, 29, 36, 43 Dasatinib Dose Level With chemoradiation Maintenance x 2 years* Dasatinib is to be taken 1x daily
  1. 50 mg daily 100 mg daily
  2. 70 mg daily 100 mg daily
  3. 100 mg daily 100 mg daily
- Group 2: Group 2: Neoadjuvant Therapy for Potentially Resectable Stage III NSCLC STUDY SCHEMA DAY Radiation 1-5 8-12 15-19 22-26 29-33 36-38 Paclitaxel 1 8 15 22 29 36 Surgery Carboplatin 1 8 15 22 29 36 Dasatinib ----------------------------------------------------------------- Maintenance Dasatinib RT: External radiotherapy 50.4 Gy, 1.8 Gy/fx for 28 fx Paclitaxel: 50 mg/m2/week over 1 hour IV infusion days 1, 8, 15, 22, 29, 36 Carboplatin: AUC = 2 IV infusion days 1, 8, 15, 22, 29, 36,
  Dasatinib Dose Level With chemoradiation Maintenance x 2 years* Dasatinib is to be taken 1x daily
  1. 50 mg daily 100 mg daily
  2. 70 mg daily 100 mg daily
  3. 100 mg daily 100 mg daily
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 11 | 0 | 11
Age, Categorical [Number; unit: participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 6 |  | 6
  >=65 years | 5 |  | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (5.38) |  | 65.5 (5.38)
Gender [Number; unit: participants]
  Female | 3 |  | 3
  Male | 8 |  | 8
Region of Enrollment [Number; unit: participants]
  United States | 11 |  | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Came Off Study for Toxicity Using CTC Version 3.0
Description: 6 patients came off study for toxicity
Time Frame: within 28 days after the last radiation treatment
Measure: Number; unit: participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 10 | 0
participants | 6 |

2. Secondary Outcome: Complete and Partial Response by CT Scan or MRI
Time Frame: within 30 days of last treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Baseline then approximately 30 days post the last dose of drug, which could be up to 2.5 years.
Groups:
- Group 1: DAY Radiation 1-5 8-12 15-19 22-26 29-33 36-40 43-47 Paclitaxel 1 8 15 22 29 36 43 Carboplatin 1 8 15 22 29 36 43 Dasatinib ----------------------------------------------------------------------Maintenance Dasatinib RT: External radiotherapy, 64.8 Gy, for 35 fx Paclitaxel: 50 mg/m2/week over 1 hour IV infusion days 1, 8, 15, 22, 29, 36, 43 Carboplatin: AUC = 2 IV infusion days 1, 8, 15, 22, 29, 36, 43 Dasatinib Dose Level With chemoradiation Maintenance x 2 years* Dasatinib is to be taken 1x daily 50 mg daily
- Group 2: DAY Radiation 1-5 8-12 15-19 22-26 29-33 36-40 43-47 Paclitaxel 1 8 15 22 29 36 43 Carboplatin 1 8 15 22 29 36 43 Dasatinib ----------------------------------------------------------------------Maintenance Dasatinib RT: External radiotherapy, 64.8 Gy, for 35 fx Paclitaxel: 50 mg/m2/week over 1 hour IV infusion days 1, 8, 15, 22, 29, 36, 43 Carboplatin: AUC = 2 IV infusion days 1, 8, 15, 22, 29, 36, 43 Dasatinib Dose Level With chemoradiation Maintenance x 2 years* Dasatinib is to be taken 1x daily
  70 mg daily
Arm/Group | Group 1 | Group 2
Serious Adverse Events (participants affected / at risk) | 2/5 | 4/5
Other Adverse Events (participants affected / at risk) | 5/5 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=5) | Group 2 (N=5)
pt #2: right leg pain (Investigations) | 1 (1) | 0 (0)
pt # 5: troponin and chest pain (4), cardiac ischemia (3), allergic reaction (2) (Investigations) | 1 (1) | 0 (0)
pt #7: hypotension, diarrhea, SVT/arrythmia (2), hypokalemia and hypomagnesmia (1) (Investigations) | 0 (0) | 1 (1)
pt #7: pleural effusion and pericardial effusion (3) (Investigations) | 0 (0) | 1 (1)
pt #8: radiation esophagitis and pain (3) (Investigations) | 0 (0) | 1 (1)
pt 10: pneumonitis/pulmonary infiltrates (4)- definitely related to Dasatinib, (Investigations) | 0 (0) | 1 (1) — f/u: death, f/u 2: death secondary to event
pt #11: infection normal ANC (penumonia) (3) (Investigations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=5) | Group 2 (N=5)
ANC (Investigations) | 2 (2) | 0 (0)
anorexia (Investigations) | 1 (1) | 1 (1)
altered eating (Investigations) | 0 (0) | 1 (1)
altered taste (Investigations) | 0 (0) | 1 (1)
anxiety (Investigations) | 0 (0) | 1 (1)
constipation (Investigations) | 1 (1) | 1 (1)
cough (Investigations) | 2 (2) | 0 (0)
dehydration (Investigations) | 0 (0) | 3 (3)
diarrhea (Investigations) | 2 (2) | 1 (1)
dyspnea (Investigations) | 1 (1) | 1 (1)
dyspepsia (Investigations) | 0 (0) | 1 (1)
dysphagia (Investigations) | 1 (1) | 3 (3)
epistaxis (Investigations) | 1 (1) | 0 (0)
esophagitis (Investigations) | 2 (2) | 2 (2)
erythema (Investigations) | 0 (0) | 1 (1)
fatigue (Investigations) | 3 (3) | 3 (3)
gynecomastis (Investigations) | 1 (1) | 0 (0)
HGB (Investigations) | 2 (2) | 0 (0)
heartburn (Investigations) | 0 (0) | 1 (1)
hoarseness (Investigations) | 1 (1) | 0 (0)
hypotension (Investigations) | 1 (1) | 0 (0)
lymphopenia (Investigations) | 4 (4) | 2 (2)
Nausea (Investigations) | 2 (2) | 3 (3)
pain (Investigations) | 1 (1) | 0 (0)
phosphorus (Investigations) | 1 (1) | 0 (0)
pleural effusion (Investigations) | 2 (2) | 0 (0)
radiation dermatitis (Investigations) | 1 (1) | 0 (0)
rash (Investigations) | 1 (1) | 0 (0)
vomiting (Investigations) | 1 (1) | 1 (1)
WBC (Investigations) | 2 (2) | 0 (0)
wt loss (Investigations) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No